CLINICAL TRIAL: NCT03668704
Title: Survivorship and Outcomes of Robotic-Arm Assisted Bicompartmental Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: St. Helena Hospital Coon Joint Replacement Institute (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2016-09-28; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; medial; bicompartmental; patellofemoral
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medial Bicompartmental Knee Arthroplasty: Patient who have received a robotic-arm assisted medial and patellofemoral knee arthroplasty.

SUMMARY:
The purpose of the study is to determine the clinical outcomes and survivorship of robotic-arm assisted medial bicompartmental knee arthroplasty at two, five, seven and ten years postoperative.

DETAILED DESCRIPTION:
The purpose of the study is to determine the survivorship, patient satisfaction and clinical outcomes of robotic-arm assisted medial bicompartmental knee arthroplasty using the MCK implant system starting at two years post-operative and continuing for five, seven and ten years post-operative.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 21 years of age who underwent robotic-arm assisted medial bicompartmental arthroplasty by the investigating surgeon and received MCK implants and are at least 24 months post-operative.
* Patient has signed an IRB approved Informed Consent Form or with IRB approved waiver of written signed consent, patient has verbally consented to study participation.
* Patient is willing to comply with follow up

Exclusion Criteria:

* Patients will be excluded from participation in the study if they are cognitively unable to answer questions related to their index procedure and health quality of life forms.
* Patient had active infection
* Implants were implanted without bone cement
* Patients did not have sufficient bone stock to allow for insertion and fixation of components
* Patient did not have sufficient soft tissue integrity to allow for stability
* Patient had a neurological or muscular deformity that did not allow for control of the knee.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 21 years of age who require a primary robotic-arm assisted medial bicompartmental arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
% of patients with Revisions | 10 years after surgery
  To determine the revision rate in this patient population

SECONDARY OUTCOMES:
% of patients with Revisions | 2 years after surgery
  To determine the revision rate in this patient population

OTHER OUTCOMES:
% of patients with revisions | 5 years after surgery
  To determine the revision rate in this patient population
% of patients with revisions | 7 years after surgery
  To determine the revision rate in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Coon, MD, Principal Investigator — St. Helena Hospital Coon Joint Replacement Institute
Locations (1):
- St. Helena Hospital Coon Joint Replacement Institute, St. Helena, California, United States

IPD SHARING:
Plan to Share IPD: No